CLINICAL TRIAL: NCT00730665
Title: A Parallel-Group, Randomized, Double-Blind, Multi-Center Dose Response Study To Evaluate The Efficacy And Safety Of PF-00885706, A 5-HT4 Receptor Partial Agonist, As Add-On Therapy To Esomeprazole For The Relief Of Symptoms In Subjects With Gastro-esophageal Reflux Disease (GERD) Who Have A Poor Response To Proton Pump Inhibitor (PPI) Treatment
Brief Title: Efficacy And Safety Of PF-00885706 For The Relief Of Symptoms In Subjects With Gastro-esophageal Reflux Disease (GERD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been placed on clinical hold by the sponsor due to operational reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A8311003
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: PPI partial responders with non-erosive GERD.
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-((4-((((3-isopropyl-2-oxo-2,3-dihydro-1H-benzimidazol-1-yl)carbonyl)amino)methyl)piperidin-1-yl)methyl)cyclobutanecarboxylic acid; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 100ug (Experimental)
  Interventions: Drug: PF-00885706; Drug: Esomeprazole
- 300ug (Experimental)
  Interventions: Drug: PF-00885706; Drug: Esomeprazole
- 1mg (Experimental)
  Interventions: Drug: PF-00885706; Drug: Esomeprazole
- 3mg (Experimental)
  Interventions: Drug: PF-00885706; Drug: Esomeprazole
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Esomeprazole

INTERVENTIONS:
Drug: PF-00885706 — Capsule, 100ug, every 12 hours (twice a day)
  Arms: 100ug
Drug: Esomeprazole — Patients entering the run-in phase lasting 6 weeks (42 days) will be switched from their current proton pump inhibitor (PPI) treatment and maintained on a standard background PPI - open label esomeprazole 20 mg to be taken once daily 1 hour before breakfast. Subjects meeting randomization criteria at Visit 4 are randomly assigned to one of the active arms of PF-00885706 or matching placebo, in addition to esomeprazole.
  Arms: 100ug
Drug: PF-00885706 — Capsule, 300ug, every 12 hours (twice a day)
  Arms: 300ug
Drug: Esomeprazole — Patients entering the run-in phase lasting 6 weeks (42 days) will be switched from their current proton pump inhibitor (PPI) treatment and maintained on a standard background PPI - open label esomeprazole 20 mg to be taken once daily 1 hour before breakfast. Subjects meeting randomization criteria at Visit 4 are randomly assigned to one of the active arms of PF-00885706 or matching placebo, in addition to esomeprazole.
  Arms: 300ug
Drug: PF-00885706 — Capsule, 1mg, every 12 hours (twice a day)
  Arms: 1mg
Drug: Esomeprazole — Patients entering the run-in phase lasting 6 weeks (42 days) will be switched from their current proton pump inhibitor (PPI) treatment and maintained on a standard background PPI - open label esomeprazole 20 mg to be taken once daily 1 hour before breakfast. Subjects meeting randomization criteria at Visit 4 are randomly assigned to one of the active arms of PF-00885706 or matching placebo, in addition to esomeprazole.
  Arms: 1mg
Drug: PF-00885706 — Capsule, 3mg, every 12 hours (twice a day)
  Arms: 3mg
Drug: Esomeprazole — Patients entering the run-in phase lasting 6 weeks (42 days) will be switched from their current proton pump inhibitor (PPI) treatment and maintained on a standard background PPI - open label esomeprazole 20 mg to be taken once daily 1 hour before breakfast. Subjects meeting randomization criteria at Visit 4 are randomly assigned to one of the active arms of PF-00885706 or matching placebo, in addition to esomeprazole.
  Arms: 3mg
Other: Placebo — Capsule, Placebo, every 12 hours (twice a day)
  Arms: Placebo
Drug: Esomeprazole — Patients entering the run-in phase lasting 6 weeks (42 days) will be switched from their current proton pump inhibitor (PPI) treatment and maintained on a standard background PPI - open label esomeprazole 20 mg to be taken once daily 1 hour before breakfast. Subjects meeting randomization criteria at Visit 4 are randomly assigned to one of the active arms of PF-00885706 or matching placebo, in addition to esomeprazole.
  Arms: Placebo

SUMMARY:
To understand the dose-response characteristics of PF-00885706 for efficacy in terms of symptomatic relief when used as add-on treatment to esomeprazole 20mg (standard proton pump inhibitor [PPI] treatment), in subjects with gastro-esophageal reflux (GERD) who have inadequate relief with PPIs.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of GERD who fulfill the following criteria:

who have symptoms for least six months prior to enrollment; who are currently on daily treatment with a PPI and have been on such treatment for at least 3 months; whose symptoms are persistent, troublesome and that include heartburn and/or regurgitation as their predominant symptoms despite treatment with a PPI; who are seeking relief of persistent symptoms.

Exclusion Criteria:

* Subjects with erosive esophagitis - An endoscopy within the last 5 years is required to verify absence.
* Subjects with any esophageal or gastric diseases/conditions that may contribute to their GERD symptoms.
* If female; pregnant, lactating or positive serum or urine pregnancy tests.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Complete resolution of heartburn and regurgitation. [i.e. no more than one day with either mild heartburn or regurgitation over the seven days prior to the assessment time-point (Visit 6 and Visit 8)] | 28 days

SECONDARY OUTCOMES:
Number of days with heartburn (daytime and night-time) | 28 days
Number of days with regurgitation (daytime and night-time) | 28 days
Number of heartburn and regurgitation-free days (24hrs) | 28 days
Composite score of heartburn and regurgitation frequency and severity | 28 days
Time to resolution of symptoms of heartburn/regurgitation | 28 days
Number of antacid rescue medication (Gaviscon) tablets used | 28 days
Severity of additional GERD symptoms | 28 days
Quality of Life (assessed using PAGI-QOL to PGIC (Patient Global Impression of Change) | 28 days
Complete resolution of heartburn | 28 days
Complete resolution of regurgitation | 28 days
Average severity of heartburn (daytime and night-time) | 28 days
Average severity of regurgitation (daytime and night-time) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Pfizer Investigational Site, Brussels, Belgium
- Brazil (4):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- France (9):
  - Pfizer Investigational Site, Nice, Cedex 3
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Laval
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Segré
  - Pfizer Investigational Site, Tours
- Germany (13):
  - Pfizer Investigational Site, Amberg
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Eisenach
  - Pfizer Investigational Site, Freising
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Koenigslutter
  - Pfizer Investigational Site, Konstanz
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Madgeburg
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Trnava
- Pfizer Investigational Site, Seoul, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8311003&StudyName=Efficacy%20And%20Safety%20Of%20PF-00885706%20For%20The%20Relief%20Of%20Symptoms%20In%20Subjects%20With%20Gastro-esophageal%20Reflux%20Disease%20%28GERD%29